CLINICAL TRIAL: NCT04341103
Title: AlloSure Guided Immuno-Optimization for COVID-19: An Early Experience
Acronym: Al-COVE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: Al-COVE
Record Dates: First submitted 2020-03-16; First posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Solid Organ Transplant Rejection; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The utilization of AlloSure to help guide immunosuppression management in solid organ transplant recipients diagnosed with COVID-19

DETAILED DESCRIPTION:
An observational case series of patients with solid organ transplants who have been admitted with suspected COVID-19 utilizing AlloSure dd-cf DNA to help guide immunosuppression management balancing the treatment of sepsis and avoiding allograft rejection.

ELIGIBILITY:
Inclusion Criteria:

* Liver, Heart, Lung or Kidney organ transplant recipient with a suspected or confirmed diagnosis of COVID-19

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Solid organ (liver, heart, lung or kidney) transplant recipients diagnosed with suspected or confirmed case of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessing the utility of AlloSure dd-cfDNA to guide clinical immune-optimization for transplant patients with COVID-19 | 6 months
  AlloSure dd-cfDNA blood draw values

IPD SHARING:
Plan to Share IPD: No